CLINICAL TRIAL: NCT05503940
Title: Association of Multiple Medications With the Severity of Dyspepsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: KY20222180-F-1
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dyspepsia is a very common gastrointestinal disease. Some medications, were associated with higher frequent incidences of dyspepsia, including non-steroid anti-inflammatory drugs (NSAIDs), Bisphosphonates, Tetracyclines, et al. Multiple medications were suggested to be strongly relate to adverse drug events (ADEs), adverse drug reactions (ADRs), drug-drug interactions, and drug-disease interactions, which may cause gastrointestinal(GI) dysfunction or injury to the GI mucosa. However, it was unclear whether multiple medications was associated with more severe symptoms of dyspepsia and dyspepsia-based score systems.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old
2. Patients who met broad criteria of dyspepsia

Exclusion Criteria:

1. organ failure defined by Marshall standard
2. severe psychiatric illnesses
3. suspected or identified bowel obstruction
4. known malignancy
5. pregnancy or lactation
6. unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years old who met broad criteria of dyspepsia were eligible for our study.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with severe dyspepsia judged by patients | 1 day
  Patients rated the severity of dyspepsia as mild, moderate, and severe by themselves

SECONDARY OUTCOMES:
Global Overall Symptom score (GOSS) | 1 days
  The GOSS consists of 10 cardinal items (epigastric pain, epigastric discomfort, Heartburn, acid regurgitation, upper abdominal bloating, belching, nausea, early satiety, postprandial fullness, other epigastric symptoms(eg. epigastric burning). Each item can be scored from 1 (no) to 7 (worst).
Functional dyspepsia | 1 days
  Functional dyspepsia was defined by Rome IV criteria. Patients diagnosed as Rome IV criteria met the following criteria: by one or more of the following symptoms: postprandial fullness, early satiation, epigastric pain, and epigastric burning that are unexplained after a routine clinical evaluation, Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.
organic upper gastrointestinal (GI) diseases. | 1 day
  All included patients underwent upper GI endoscopy and abdominal ultrasound and H. Pylori test. Barrett's esophagus, esophageal candidiasis, esophageal cancer, gastric ulcer, gastric erosion, gastric cancer, duodenal ulcer, duodenal erosion, cholecystitis, pancreatitis and biliary stones were classified as organic upper GI diseases.
subtypes of functional dyspepsia | 6 months
  functional dyspepsia was classified into three subgroups：(1) Postprandial Distress Syndrome, defined as Bothersome postprandial fullness or/and Bothersome early satiation. (2) Bothersome epigastric pain AND/OR Bothersome epigastric burning. (3) mixed syndrome, defined when postprandial distress syndrome and epigastric pain syndrome presented simultaneously.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1 day
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hospital anxiety and depression scale | 1 day
  Anxiety and depression of patients are assessed by using Hospital Anxiety and Depression Scale.It contains 14 items (7 anxiety and 7 depression), which assess symptoms experienced during the past week on a 0-3 scale. A subscore of > 8 for depression or anxiety would indicate a clinical case.
Quality of Life scores | 1 day
  Quality of Life scores assessed by Patient-reported outcomes measurement information system (PROMIS) Global-10 questionnaire.PROMIS Global-10 is a newly validated 10-question survey used to assess health care-related quality of life measures for the general population.
  It's a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient and a better quality of life.
Number of Participants with other functional gastrointestinal diseases | 1 day
  Other functional gastrointestinal diseases，such as irritable bowel syndrome(IBS) or functional heartburn，etc.
Functional dyspepsia symptom diary (FDSD) score | 1 days
  The FDSD consists of 5 cardinal items (burning in the stomach, stomach pain, bloating, postprandial fullness, and early satiety) and 3 supplementary items (nausea, burping/belching rating, and burping/belching bother). Each item can be scored from 0 (no) to 10 (worst). Total Symptom Score includes the 5 cardinal items and ranges from 0 to 50

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing 986 Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi